CLINICAL TRIAL: NCT05436639
Title: SPI-62 as a Treatment for Hypercortisolism Related to a Benign Adrenal Tumor
Acronym: ACSPIRE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data does not demonstrate a clear benefit for this patient population, and we therefore cannot justify continuing this trial.
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-62-CL-2002
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-05

CONDITIONS: Autonomous Cortisol Secretion (ACS); ACTH-Independent Cushing Syndrome; ACTH-Independent Adrenal Cushing Syndrome, Somatic
Keywords: Autonomous Cortisol secretion (ACS); ACTH-independent adrenal Cushing's syndrome (aCs); benign adrenal tumor
MeSH Terms: conditions — Acth-Independent Macronodular Adrenal Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SPI-62 dose (Experimental): 2mg dose level of SPI-62. Active drug by mouth.
  Interventions: Drug: SPI-62 dose

INTERVENTIONS:
Drug: SPI-62 dose — SPI-62 is an 11β hydroxysteroid dehydrogenase type 1 (HSD-1) inhibitor, supplied as oral tablets for dose 2 of drug (2mg).

SUMMARY:
This is study with SPI-62 to evaluate the efficacy, safety, and pharmacological effect of SPI-62 in subjects with hypercortisolism related to a benign adrenal tumor. Each subject will receive 2mg of SPI-62 daily.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm study, Phase 2 study to estimate SPI-62's effect on clinical features of hypercortisolism related to a benign adrenal tumor, including diabetes/impaired glucose tolerance, hyperlipidemia, hypertension, and osteopenia. Each subject who provides consent and meets all inclusion and exclusion criteria will participate in a screening period and an open-ended treatment period. Visits occur at screening/baseline, months 1, 3, 6, 9, and 12, and then quarter-annually.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis and main criteria for inclusion and exclusion:

The following are the main inclusion criteria:

* Adults able to provide informed consent.
* Documented characteristically benign adrenal nodule, with diameter ≤ 4 cm, homogenous texture, and non-contrast computerized tomography ≤ 20 HU attenuation or proven to be non malignant.
* Diagnosis of diabetes mellitus, pre-diabetes or impaired glucose tolerance, either untreated or on stable standard of care treatment, based on at least one of:

  * HbA1c ≥ 5.7% but not > 9.5%
  * 2-hour glucose level ≥ 7.8 mmol (140 mg/dL) on a 75 g OGTT
* At least one additional documented cortisol-related morbidities, either untreated or on stable standard of care treatment:

  * hypercholesterolemia with total cholesterol > 3.9 mM (150 mg/dL);
  * hypertriglyceridemia with triglycerides > 2.3 mM (200 mg/dL);
  * osteopenia with bone densitometry Z-score < -2.0 or T-score < -1.0;
  * history or evidence of minimally traumatic or osteoporotic fracture; or
  * hypertension with resting supine blood pressure > 130 but < 180 mmHg systolic or > 85 but < 120 mmHg diastolic.
* Poorly suppressible hypercortisolemia:

  * Morning serum cortisol > 50 nM (1.8 mcg/dL) after a 1 mg ONDST.
  * Subjects with dexamethasone < 3.3 nmol/L (130 ng/dL) will undergo a high-dose (8 mg) ONDST.
  * Subjects who take estrogen-containing medicines will be evaluated based on free cortisol > 2.2 nM (80 ng/dL).
  * For subjects with morning serum cortisol > 138 nM (5.0 mcg/dL) after ONDST, the Investigator will assess for adrenal Cushing's syndrome.

Exclusion Criteria:

* Diagnosis of ACTH-dependent Cushing's syndrome, pheochromocytoma, aldosteronoma, adrenocortical carcinoma, or congenital adrenal hyperplasia, or other malignancy associated hypercortisolism including history of adrenal carcinoma.
* History of adrenalectomy or planned adrenalectomy within 4 months after randomization.
* Exogenous hypercortisolism.
* Uncontrolled, clinically significant hypo- or hyperthyroidism.
* History of idiopathic thrombocytopenia.
* Moderately impaired renal function (estimated glomerular filtration rate < 60 mL/min/1.73m2).
* History of cancer (other than non-melanoma skin, thyroid, or early-stage prostate cancer) within 3 years.
* Any major surgery, or significant post-operative sequelae, within 1 month prior to informed consent or planned during the trial.
* Pregnant or lactating.
* Positive test for severe acute respiratory syndrome coronavirus 2 infection within 4 weeks, or hospitalization for Coronavirus disease 2019 within 6 months, prior to randomization.
* Any other current or prior medical condition expected to interfere with the conduct of the trial or the evaluation of its results.
* Participation in any clinical trial within 3 months prior to the first dose of study drug, or longer depending on half-life of the investigational therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c at Week 6 | Baseline to week 6
  HbA1c change from baseline
Change in HbA1c at week 12 | Baseline to week 12
  HbA1c change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, MD, Study Chair — Sparrow Pharmaceuticals
Locations (5):
- United States (2):
  - Mayo Clinic Cancer Center (MCCC) - Rochester, Rochester, Minnesota
  - Ohio State McCampbell Outpatient Care, Columbus, Ohio
- Romania (2):
  - C.M.D.T.A. Neomed, Brasov
  - Institutul National de Endocrinologie, Bucharest
- King's College Hospital, London, United Kingdom